CLINICAL TRIAL: NCT00699543
Title: The Efficacies of The New Paclitaxel-Eluting CoroflexTM Please Stent in Percutaneous Coronary Intervention: Comparison or Efficacy Between COroflex PLEASe ANd TaxusTM Stent
Brief Title: The Efficacies of The New Paclitaxel-Eluting CoroflexTM Please Stent in Percutaneous Coronary Intervention
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Hyo-Soo, Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECO-PLEASANT
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C (Experimental): Coroflex Please stent implantation
  Interventions: Device: Coroflex Please stent implantation
- T (Active Comparator): Taxus stent implantation
  Interventions: Device: Taxus stent implantation

INTERVENTIONS:
Device: Coroflex Please stent implantation — Use Coroflex Please stent in the treatment of coronary stenosis
  Other Names: Coroflex Please stent
  Arms: C
Device: Taxus stent implantation — Use Taxus stent in the treatment of coronary stenosis
  Other Names: Taxus stent
  Arms: T

SUMMARY:
Objectives

: To evaluate the clinical efficacy, angiographic outcomes, and safety of the new paclitaxel-eluting coronary stent (CoroflexTM Please, B Braun, Germany), compared with another paclitaxel-eluting coronary stent system (TaxusTM, Boston Scientific, USA) in the treatment of coronary stenosis.

Study Design

: Prospective, open label, 2: 1 randomized multi-center trial. Patients will be randomized according to the type of drug eluting stent ( CoroflexTM Please vs. TaxusTM). Randomization will also be stratified per hospital for the presence of DM and the presence of long lesions (lesion length > 28mm)

Patient Enrollment

:915 patients enrolled at 13 centers in Korea.

Patient Follow-Up

:Clinical follow-up will occur at 1, 4, 9, 12 months and 2, 3years after intervention. Investigator or designee may conduct follow-up as telephone contacts or office visits.

Primary Endpoint

:Clinically driven Target vessel Revascularization (TVR) at 9 months.

Secondary Endpoints

:A. Clinical safety and efficacy end points

1. Major Cardiac Adverse Events (MACE; All Death, cardiac death, Myocardial infarction (Q-wave and non-Q wave), TVR)
2. Target Vessel Failure (TVF; cardiovascular death, myocardial infarction, clinically driven TVR)
3. Stent thrombosis

B. Angiographic efficacy end points

1. in-stent binary restenosis by QCA
2. in-stent and in-lesion late loss by QCA
3. in-stent and in-lesion MLD and percentage diameter stenosis by QCA immediately after the index procedure and at 9 months of follow-up

ELIGIBILITY:
Inclusion Criteria

* General Inclusion Criteria

  1. Subject must be at least 18 years of age.
  2. Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving the CoroflexTM Please stent and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
  3. Subject must have coronary artery stenosis (>50% by visual estimate) with evidence of myocardial ischemia (e.g., stable, unstable angina, myocardial infarction, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia.) or Subject must have significant coronary artery stenosis (>70% by visual estimate)
* Angiographic Inclusion Criteria

  1. Target lesion(s) must be located in a native coronary artery with visually estimated diameter of ≥ 2.5 mm and ≤ 4.0 mm.
  2. Target lesion(s) must be amenable for percutaneous coronary intervention

Exclusion Criteria

* General Exclusion Criteria

  1. The patient has a known hypersensitivity or contraindication to any of the following medications:

     * Heparin
     * Aspirin
     * Both Clopidogrel and Ticlopidine
     * Paclitaxel
     * Stainless steel
     * Contrast media(*) (*)Patients with documented sensitivity to contrast media which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.
  2. Systemic (intravenous) Paclitaxel use within 12 months.
  3. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
  4. History of bleeding diathesis or known coagulopathy (including heparin- induced thrombocytopenia), or will refuse blood transfusions.
  5. Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
  6. An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 6 months post enrollment.
  7. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
  8. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
  9. Patients with LVEF<25% or those with cardiogenic shock
  10. Patients with acute ST elevation myocardial infarction who requires primary PCI
  11. Patients with acute ST elevation myocardial infarction within 48hrs
  12. Creatinine level ≥ 3.0mg/dL or dependence on dialysis.
* Angiographic Exclusion Criteria

  1. Patients with significant left main stem stenosis which requires revascularization therapy
  2. Patients who's target lesion has in-stent restenosis at the stented segment of drug-eluting stents or bare metal stents
  3. Target lesions with bifurcating disease which require side branch stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Estimated)
Dates: Start 2008-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Clinically driven Target vessel Revascularization (TVR) | 9 months.

SECONDARY OUTCOMES:
Major Cardiac Adverse Events (MACE; All Death, cardiac death, Myocardial infarction (Q-wave and non-Q wave), TVR) | 1, 4, 9, 12 months and 2, 3years
Target Vessel Failure (TVF; cardiovascular death, myocardial infarction, clinically driven TVR) | 1, 4, 9, 12 months and 2, 3years
Stent thrombosis | 1, 4, 9, 12 months and 2, 3years
In-stent binary restenosis by QCA | 9 months
In-stent and in-lesion late loss by QCA | 9 months
In-stent and in-lesion MLD and percentage diameter stenosis by QCA | Immediately after the index procedure and at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital; In-Ho Chae, MD, PhD, Study Chair — Seoul National University Bundang Hospital; Seung-Ho Hur, MD, Ph, Study Chair — Keimyung University Dongsan Medical Center; Tae-Jin Youn, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital; Soo-Joong Kim, MD, PhD, Principal Investigator — Kyunghee University Medical Center; Keum-Soo Park, MD, PhD, Principal Investigator — Inha University Hospital; Byung-Ok Kim, MD, PhD, Principal Investigator — Inje University Sang-gye Paik Hospital; Min-Su Hyon, MD, PhD, Principal Investigator — Soon Chun Hyang University Hospital; Sang-Wook Kim, MD, PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Jong-Seon Park, MD, PhD, Principal Investigator — Yeungnam University Hospital; Doo-Il Kim, MD, PhD, Principal Investigator — Inje University; Tae-Joon Cha, MD, PhD, Principal Investigator — Kosin University Gospel Hospital; Sang-Gon Lee, MD, PhD, Principal Investigator — Ulsan University Hospital; Hee-Kyoung Jeon, MD, PhD, Principal Investigator — Uijeongbu St. Mary's Hospital

REFERENCES:
- [Derived] Seo JB, Kang SH, Hur SH, Park KW, Youn TJ, Park JS, Yang HM, Lee HY, Kang HJ, Koo BK, Bae JH, Kim SW, Moon KW, Choi JW, Lee SG, Chung WY, Kim SJ, Kim DI, Kim BO, Hyon MS, Park KS, Cha TJ, Yoo CW, Jeon HK, Kim HS. Randomized trial comparing the efficacy between different types of paclitaxel-eluting stents: the comparison of efficacy between COroflex PLEASe ANd Taxus stent (ECO-PLEASANT) randomized controlled trial. Am Heart J. 2013 May;165(5):733-43. doi: 10.1016/j.ahj.2013.02.009. Epub 2013 Mar 20. PMID 23622910
- [Derived] Seo JB, Jeon HK, Park KW, Park JS, Bae JH, Kim SW, Moon KW, Choi JW, Lee SG, Chung WY, Youn TJ, Kim SJ, Kim DI, Kim BO, Hyon MS, Park KS, Cha TJ, Hwang HK, Hur SH, Kim HS. Efficacies of the new paclitaxel-eluting Coroflex Please stent in percutaneous coronary intervention; comparison of efficacy between Coroflex Please and Taxus (ECO-PLEASANT) trial: study rationale and design. Trials. 2009 Oct 23;10:98. doi: 10.1186/1745-6215-10-98. PMID 19849864